CLINICAL TRIAL: NCT03131427
Title: A Nation-wide Hospital-based Registry:China Registry for Genetic / Metabolic Liver Diseases
Brief Title: China Registry for Genetic / Metabolic Liver Diseases
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing YouAn Hospital (Other); Henan Provincial People's Hospital (Other); Beijing Ditan Hospital (Other); Hebei Medical University Third Hospital (Other); Peking University First Hospital (Other); Xinjiang Uygur Autonomous Region Traditional Chinese Medicine Hospital (Unknown); Nanfang Hospital, Southern Medical University (Other); Logistics University of Chinese People's Armed Police Forces (Other); Beijing Anzhen Hospital (Other); West China Second University Hospital (Other); Jinshan Hospital Fudan University (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Jidong Jia, Liver Research Center, Beijing Friendship Hospital
Other Study IDs: CR-GMLD
Record Dates: First submitted 2017-04-21; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Genetic/Metabolic Liver Diseases
Keywords: Wilson's Disease; Hereditary Hemochromatosis; Hereditary Hyperbilirubinemias; Inherited Cholestatic Liver Disease; Genetic Testing
MeSH Terms: conditions — Hepatolenticular Degeneration; Hemochromatosis; Hyperbilirubinemia, Hereditary | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Wilson's Disease: Patients who were diagnosed or possibly diagnosed with Wilson's disease. The diagnosis can be made or possibly made on the basis of Wilson's disease scoring system proposed by the Working Party at the 8th International Meeting on Wilson's disease, Leipzig 2001.
  Interventions: Drug: Standard of care
- Hereditary Hemochromatosis: Hereditary hemochromatosis can be clinically diagnosed if: ① transferrin saturation≥45% and/or elevated ferritin; ② iron overload in liver and/or spleen on magnetic resonance imaging (MRI) of liver or on liver histology; ③ exclude causes of secondary iron overload, such as alcoholic or other chronic liver disease, iron-overloading anemia, and parenteral iron overload.
  Interventions: Drug: Standard of care
- Hereditary Hyperbilirubinemias: Hereditary hyperbilirubinemias involve four syndromes: Gilbert, Crigler-Najjar, Dubin-Johnson and Rotor, among which the first two are characterized by unconjugated hyperbilirubinemia and the second two by conjugated hyperbilirubinemia. Diagnosis of hereditary hyperbilirubinemia should exclude other causes of hyperbilirubinemia, such as obstructive bile duct (slerosing cholangitis, calculi, parasites), intrahepatic cholestasis(drugs, hepatitis, immune-mediated, infectious), acute or chronic hepatocellular injury(sepsis, parenteral nutrition, severe blood loss/hypotension, trauma, conjestive heart failure), increased bilirubin production(hemolysis, hematological disease), decreased bilirubin uptake (drugs, portosystemic shunting ), reduced conjugation activity (neonatal, thyroid disease, chronic hepatitis/inflammation, wilson's disease).
  Interventions: Drug: Standard of care
- Inherited Cholestatic Liver Disease: Patients who were diagnosed or possibly diagnosed with Inherited cholestatic liver disease, including progressive familial intrahepatic cholestasis(PFIC) and benign recurrent intrahepatic cholestasis(BRIC).
  Interventions: Drug: Standard of care
- Other genetic/metabolic liver diseases: Patients who were diagnosed or possibly diagnosed with genetic/metabolic liver diseases except for Wilson's disease, hereditary hemochromatosis, hereditary hyperbilirubinemias or inherited cholestatic liver disease.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Standard of care — Standard of care according to the updated national and/or international guidelines

SUMMARY:
CR-GMLD registry started on June 13, 2015 to collect cases of genetic/metabolic liver diseases from tertiary or secondary hospitals in mainland China. Demographics, diagnosis, laboratory test results, family history and prescriptions were recorded. Patients' whole blood and serum were collected for genetic testing and future researches. These patients will be followed-up every six to twelve months.

DETAILED DESCRIPTION:
This web-based database was launched on June 13, 2015 and consists of tertiary or secondary hospitals with special interest and expertise on managing genetic/metabolic liver diseases patients across mainland China. The main inclusion criteria for this registration are patients who were diagnosed or possibly diagnosed with Wilson's disease, hereditary hemochromatosis, hereditary hyperbilirubinemias, inherited cholestatic liver disease or other genetic/metabolic liver diseases. At the first time of data entry, demographics, medical history, biochemistry and hematology results, radiology reports, diagnosis and treatment information were recorded. Patients' whole blood and serum were collected for molecular genetic testing and future researches. Then the registered patients will receive standard of care and be followed-up every 6 to 12 months. On each visit, biochemical, radiological reports, as well as clinical progress were recorded.

ELIGIBILITY:
Inclusion Criteria:

Patients who were diagnosed or possibly diagnosed with Wilson's disease, hereditary hemochromatosis, hereditary hyperbilirubinemias, inherited cholestatic liver disease or other genetic/metabolic liver diseases.

Exclusion Criteria:

Patients who are unable or unwilling to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry is a multicenter and observational study enrolling patients with genetic/metabolic liver disease across mailand China.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-06-13 (Actual); Primary Completion 2022-04-28 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
rate of liver-related events of each disease. | 10 years
  Rates of cirrhosis, decompensation and hepatocellular carcinoma.

SECONDARY OUTCOMES:
Genotype profile in Chinese patients of each disease | 10 years
Natural history of Chinese patients with each disease of different genotype | 10 years
Causes of death in Chinese patients of each disease | 10 years

OTHER OUTCOMES:
Quality of life | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jidong Jia, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (12):
- China (12):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Henan Provincial Hospital, Zhengzhou, Henan
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Jinshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Women's and Children's Hospital, Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital, Logistics University of People's Armed Police Force, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Autonomous Region Traditional Chinese Medicine Hospital, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu A, Lv T, Zhang B, Zhang W, Ou X, Huang J. Development and evaluation of an unlabeled probe high-resolution melting assay for detection of ATP7B mutations in Wilson's disease. J Clin Lab Anal. 2017 Jul;31(4):e22064. doi: 10.1002/jcla.22064. Epub 2016 Sep 17. PMID 27638368
- [Background] Lv T, Li X, Zhang W, Zhao X, Ou X, Huang J. Recent advance in the molecular genetics of Wilson disease and hereditary hemochromatosis. Eur J Med Genet. 2016 Oct;59(10):532-9. doi: 10.1016/j.ejmg.2016.08.011. Epub 2016 Aug 31. PMID 27592149
- [Derived] Zhang W, Li Y, Xu A, Ouyang Q, Wu L, Zhou D, Wu L, Zhang B, Zhao X, Wang Y, Wang X, Duan W, Wang Q, You H, Huang J, Ou X, Jia J; China Registry of Genetic/Metabolic Liver Diseases (CR-GMLD) Group. Identification of novel non-HFE mutations in Chinese patients with hereditary hemochromatosis. Orphanet J Rare Dis. 2022 Jun 6;17(1):216. doi: 10.1186/s13023-022-02349-y. PMID 35668470